CLINICAL TRIAL: NCT05858957
Title: The Effect of Magnesium Sulfate on Extubation Quality Score and Recovery in Larynx Laser Microsurgery, Prospective, Randomized, Controlled Study
Brief Title: Magnesium Sulphate and Extubation Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Associate professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Extubation quality
Record Dates: First submitted 2023-04-18; First posted 2023-05-15 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-04

CONDITIONS: Perioperative Complication
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium (Experimental): Magnesium sulfate 30 mg/kg with 100 ml saline will apply in 10 min before induction of general anesthesia (maximum magnesium dose 2g) (Group M) . When the magnesium infusion completed, general anesthesia induction will start.
  Interventions: Drug: Magnesium sulfate
- Saline (Active Comparator): saline 100 ml will apply in 10 min before induction of general anesthesia (Group S) . When the saline infusion completed, general anesthesia induction will start.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Magnesium sulfate — magnesium sulphate IV 30 mg/kg (10 min) infusion apply to the Group M
  Other Names: Intravenous magnesium infusion
  Arms: Magnesium
Drug: Saline — 100 ml saline infusion apply to the Group S
  Other Names: Saline infusion
  Arms: Saline

SUMMARY:
The investigators aimed to search effect of magnesium Sulfate on extubation quality scores, recovery and pain in larynx micro surgery. The patients allocated to two groups to receive magnesium sulfate 30 mg/kg in 100 ml saline infusion (maximum 2g) (Group m) or saline 100 ml (Group S) before induction of anesthesia. Anesthesia induction performed with propofol 2 mg/kg, rocuronium 0.6 mg/kg, remifentanil 0.5 µg/kg and general anesthesia maintained with total intravenous anesthesia (propofol 3-7 mg/kg, remifentanil 0.05-0.1 µg/kg/min and O2/air 30/70 mixture) to the all patients. Extubation quality scores, Extubation time, NRS scores were assessed.

DETAILED DESCRIPTION:
The investigators aimed to search effect of magnesium sulfate on extubation quality, recovery feature and complications.98 adult patients scheduled for larynx laser microsurgery were included and randomly allocated to two groups to receive magnesium sulfate 30 mg/kg in 100 ml saline infusion (maximum 2g) (Group m) or saline 100 ml (Group S) before induction of anesthesia. Anesthesia induction performed with propofol 2 mg/kg, rocuronium 0.6 mg/kg, remifentanil 0.5 µg/kg and general anesthesia maintained with total intravenous anesthesia (propofol 3-7 mg/kg, remifentanil 0.05-0.1 µg/kg/min and O2/air 30/70 mixture) to the all patients. Paracetamol 15 mg/kg applied to all patients.Extubation quality score, extubation time, stay in postanesthesia unit (PACU) time, numeric rating scale (NRS) and complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18 age over
* American society of Anesthesiology (ASA) clinical status I-III
* the patients who experience larynx micro surgery

Exclusion Criteria:

* under 18 years old
* ASA IV and over
* severe airway obstruction
* neuromuscular disease
* presence of tracheostomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
extubation quality scores | at the time between stop the total intravenous anesthesia and extubation of patient (last 20 min of anesthesia).
  Extubation quality will assess with quality scores such as no cough, Mild cough, moderate cough, severe cough.

SECONDARY OUTCOMES:
extubation time | time between stop the total intravenous anesthesia and extubation of patient (last 20 min of anesthesia).
  The time need to adequate spontaneous ventilation at recovery period

CONTACTS AND LOCATIONS:
Overall Officials: ebru biricik, Principal Investigator — çukurova university faculty of medicine
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No